CLINICAL TRIAL: NCT02832908
Title: Evaluation of the Physiopathological Phenomena and the Haemodynamic and Cerebral Metabolic Effects From Semi-seated Position to Lying Position in Patients With Brain Trauma
Acronym: PULSATILITY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9413
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients + parents (Other): Patients with severe head trauma
  Interventions: Other: Change from semi-seated position to supine

INTERVENTIONS:
Other: Change from semi-seated position to supine — from semi-seated position (30°) to lying position

SUMMARY:
Brain trauma is an important burden in traumatologic intensive care. In these patients the treatment is guided by a cluster of multimodal monitoring parameters. Despite this it is difficult to assess the actual physiopathologic status of the brain. Changing the position of these patients (semi-seated to lying position) causes changes in the hémodynamics brain conditions, so in monitoring parameters . The analysis of these changes can givr us valuable clinically informations.

DETAILED DESCRIPTION:
Severe brain trauma (CGS < 8 ) are included. PIC, PA, PVC, EKG, airway pressure, SjO2 and NIRSS are continuously monitored.

The patients are in semi seated (30°) position. Once a day they are in supine (0°) for 30 minutes. We record every parameters before and at the end of this supine period.

After time domain and frequency domain signal processing, this parameters are compared to deduct clinical relevant conclusions.

ELIGIBILITY:
Inclusion Criteria:

* patients with a severe head trauma estimated by the Glasgow Coma Scale and by the Glasgow Outcome Scale
* age > 18

Exclusion Criteria:

* Other neurological pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
ASSESSMENT OF THE CEREBRAL OXYGENATION | UP TO 6 MONTHS

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lapeyronie - Département Anesthésie Réanimation A, Montpellier, France

REFERENCES:
- [Derived] Dagod G, Roustan JP, Bringuier-Branchereau S, Ridolfo J, Martinez O, Capdevila X, Charbit J. Effect of a temporary lying position on cerebral hemodynamic and cerebral oxygenation parameters in patients with severe brain trauma. Acta Neurochir (Wien). 2021 Sep;163(9):2595-2602. doi: 10.1007/s00701-021-04851-x. Epub 2021 Jul 8. PMID 34236525